CLINICAL TRIAL: NCT03110718
Title: Can Upper Limb Robotic Rehabilitation Plus Muscle Vibration Improve Motor Function? A Pilot Study
Brief Title: Role of Armeo-Power and Muscle Vibration in Upper Limb Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Principal investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42/2013
Record Dates: First submitted 2017-04-01; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: robotic rehabilitation; muscle vibration; combined approach
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ArmeoP+real MV (Experimental): The patients underwent forty 1h Armeo-P training sessions (i.e. five times a week for eight consecutive weeks). During the first session, the device was adjusted to the patient's arm size and the angle of suspension. The working space and the exercises were selected once the UL had been fitted with the system. All the subjects in the arm received a focal belly-muscle vibration on the spastic antagonist muscles (i.e. triceps brachialis-TB, deltoid-DE, and supraspinatus-SS) during shoulder abduction and elbow extension. MV was delivered by a pneumatic vibrator powered by compressed air, wired to appropriate-muscle probe diameter (up to 2cm2). MV was set at a frequency of 80Hz and an individually adjusted vibration amplitude so that it was just below the threshold for perceiving an illusory movement. The investigators chose such set up to avoid any signs of muscle contraction potentially reflecting either possible voluntary movement or occurrence of the tonic vibration reflex (TVR).
  Interventions: Device: ArmeoP+real MV
- ArmeoP+ Sham MV (Active Comparator): The patients underwent the same Armeo-P trainingas the experimental group. Only the vibration protocol was didderent. Indeed, in the control group a sham vibration was used, while in the experimental group, patients underwent a real one.
  Sham vibration was delivered to the control group using the same procedure of the experimental group;however, vibration intensity was subthreshold (i.e. 50mBar below the threshold).
  Interventions: Device: ArmeoP+real MV

INTERVENTIONS:
Device: ArmeoP+real MV — All the subjects assigned to the experimental received a focal belly-muscle vibration on the spastic antagonist muscles (i.e. triceps brachialis-TB, deltoid-DE, and supraspinatus-SS) during shoulder abduction and elbow extension. MV was delivered by a pneumatic vibrator powered by compressed air (Vibraplus; @Circle, San Pietro in Casale, Italy) (fig. 2) wired to appropriate-muscle probe diameter (up to 2cm2). MV was set at a frequency of 80Hz and an individually adjusted vibration amplitude (approximately 2mm in indentation depth, mean pressure of 250mBar, which effectively induce inhibition of the monosynaptic reflex) so that it was just below the threshold for perceiving an illusory movement. We chose such set up to avoid any signs of muscle contraction potentially reflecting either possible voluntary movement or occurrence of the tonic vibration reflex (TVR).

SUMMARY:
Muscle vibration (MV) has been suggested as a useful non-pharmacological approach to control spasticity. Armeo Power® (AP) is a robotic exoskeleton for rehabilitation allowing early rehabilitation treatment. The objective of our study was to determine whether AP training coupled with MV applied on antagonist muscles of the spastic upper limb (UL) can reduce the spasticity of agonist muscles. We enrolled 20 chronic post-stroke patients, who underwent 40 daily sessions of AP training. Ten subjects (group-A) received muscle MV (on triceps brachii, deltoid, and supraspinatus), whereas the other 10 (group-B) underwent a sham vibration.

ELIGIBILITY:
Inclusion Criteria:

* a first ever supra-tentorial unilateral (left hemisphere) ischemic stroke experienced more than three months before the enrollment;
* a deficit of shoulder abductor, arm flexor, and elbow extensor muscles ranging from 2 to 4 on the Medical Research Council scale (MRC);
* a spasticity of biceps brachii (BB), pectoralis major (PM), and latissimus dorsi (LD) (namely, spastic agonist muscles) ranging from 1+ to 3 on the Modified Ashworth Scale (MAS);
* age between 50 and 80 years; and (v) Caucasian ethnicity.

Exclusion Criteria:

* history of concomitant neurodegenerative diseases or brain surgery;
* severe cognitive (Mini-Mental State Examination score <23 points) or language impairment (Boston Disability Aphasia Quotient <4/5);
* severe neglect (Catherine Bergego Scale >15/30);
* systemic, bone, or joint disorders, tumors, changes in either central or peripheral sensitivity as well as visual impairments able to interfere with the aims and methods of the research;.(v) concomitant use of drugs for spasticity;
* botulin toxin treatment in the last eight months;.(vii) TMS contraindications;
* history of psychosis;
* limited passive range of motion (shoulder abduction <60°, elbow extension <30°, specified by a goniometric assessment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of spasticity-MAS | Six months
  The primary outcomes consisted in the effects of MV and Armeo Power® on spasticity by a clinical (MAS from spastic agonist muscles causing arm adduction, inward rotation, and flexion, and forearm flexion)

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of UL motor recovery after stroke -FMA | Six months
  The investigators measured the effects of MV and Armeo Power® on UL motor function impairment (measured by Fugl-Meyer Assessment of UL motor recovery after stroke -FMA).